CLINICAL TRIAL: NCT06103435
Title: Multivisceral Resections for Locally Advanced Gastric Cancer
Acronym: TOCCATA
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Marek Sierzega, Professor, Jagiellonian University
Other Study IDs: GC_MVR
Record Dates: First submitted 2023-10-18; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; locally advanced cancers; multivisceral resections; splenectomy; pancreatectomy; colectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Extent od surgical resection

SUMMARY:
The goal of this observational study is to assess whether the postoperative course and survival of patients subject to multivisceral resections for locally advanced gastric cancer (cT4b) were affected by the extent of surgery. An electronic database of 1476 patients with non-metastatic gastric cancer treated between January 1996 and December 2020 will be reviewed. The main questions it aims to answer are:

* Does splenectomy, distal pancreatectomy or partial colectomy affect postoperative complications
* What factors affect prognosis of patients with locally advanced gastric cancer

ELIGIBILITY:
Inclusion Criteria:

* gastric adenocarcinoma
* intraoperatively suspected infiltration of surrounding organs (stage cT4bN0-3bM0)
* partial or total gastrectomy

Exclusion Criteria:

* distant metastases (M1)
* gastrectomy combined with resection of organs other than spleen, pancreas, or colon

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with resectable gastric cancer treated between January 1996 and December 2020 in the First Department of Surgery, Jagiellonian University Medical College
Sampling Method: Non-Probability Sample
Enrollment: 1476 (Actual)
Dates: Start 1996-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Complications | up to 90 days
  Type and severity of complications graded by Clavien-Dindo scoring system (from 0 to 5, higher scores mean worse outcome)
Survival | Overall survival from surgery to death or last follow up, whichever came first, assessed up to 60 months
  Overall survival

SECONDARY OUTCOMES:
Rate of reoperations | up to 90 days
  Reoperations
Length of postoperative hospital stay | Up to 6 months
  Hospital stay
Rate of readmissions | One year from surgery
  Readmission

CONTACTS AND LOCATIONS:
Overall Officials: Marek Sierżęga, MD, PhD, Principal Investigator — Jagiellonian University
Locations (1):
- First Department of Surgery, Jagiellonian University Medical College, Krakow, Małopolska, Poland